CLINICAL TRIAL: NCT06844812
Title: The Effect of Methylphenidate Treatment on Oxidative Stress Levels in Children Diagnosed With Attention Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Enes Faruk ALTUNKILIÇ, Principal Investigator, Saglik Bilimleri Universitesi
Other Study IDs: 2024-05-27
Record Dates: First submitted 2025-02-15; First posted 2025-02-25 (Actual); Results first posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
Keywords: methylphenidate; Attention Deficit Hyperactivity Disorder; ADHD; oxidative stress
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples Without DNA — serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient group: Patient group with attention deficit and hyperactivity disorder. The group planned to start methylphenidate treatment independent of the study
  Interventions: Other: This is not an interventional study. Patients who are planned to start methylphenidate treatment have been invited to participate in the study.

INTERVENTIONS:
Other: This is not an interventional study. Patients who are planned to start methylphenidate treatment have been invited to participate in the study. — This is not an interventional study. Patients diagnosed with Attention Deficit Hyperactivity Disorder (ADHD), for whom methylphenidate treatment is planned, have been invited to participate in the study. The patients have been enrolled in follow-up, and our contact information has been provided to them. As part of routine care, patients have been called in once a month. Necessary dosage adjustments have been made in accordance with medical guidelines, without any intervention for the study. Patients with complaints or those who needed to be seen earlier have been seen in between. As a result, the patients were followed for a total of 3 months for this study. Serum samples for oxidative stress markers were collected at baseline (before treatment started) and at the 3rd month (after treatment began).
  Other Names: methylphenidate; ADHD treatment

SUMMARY:
The aim of this study is to investigate the effect of methylphenidate treatment on oxidative stress by measuring the levels of Total Oxidant Status (TOS), Total Antioxidant Status (TAS), Oxidative Stress Index (OSI=TOS/TAS), Malondialdehyde (MDA), Oxidized LDL (Ox-LDL), and Superoxide Dismutase (SOD) in serum samples of patients diagnosed with Attention Deficit Hyperactivity Disorder (ADHD) who have either started or are planned to start methylphenidate treatment. The measurements will be taken at baseline (0 months, before treatment initiation) and at the 3rd month (after treatment has begun) to assess the effect of methylphenidate on oxidative stress. Patients who were already planned to begin methylphenidate treatment will be invited to participate in this study. Since this is not an interventional study, no additional treatments will be administered or altered beyond the treatment the patient is already required to receive.

DETAILED DESCRIPTION:
The study population will consist of patients who are diagnosed with "Attention Deficit Hyperactivity Disorder (ADHD)" according to DSM-5-TR, who have applied to the child and adolescent psychiatry outpatient clinics of Bakırköy Prof. Dr. Mazhar Osman Mental Health and Neurological Diseases Training and Research Hospital and have been started or planned to start methylphenidate treatment by the physician they have been examined by. After an in-clinic announcement, these patients will be directed to the researcher, Enes Faruk Altunkılıç. After being informed both verbally and in writing through the informed consent process, those who agree to participate, sign the informed consent form, and meet the inclusion and exclusion criteria will be included in the study. It will also be explained to the patients and their families that their participation or non-participation in this study will not affect the treatment they will receive.

After informed consent, a structured clinical interview for DSM-5-TR will be conducted using the "Mood Disorders and Schizophrenia Form for School-Aged Children - Now and Lifetime DSM-5 - Turkish Adaptation (ÇDŞG-ŞY-DSM-5-T)." To obtain sociodemographic and clinical data for the participants, the "Sociodemographic and Clinical Data Form" created by the researchers will be completed. For the ADHD diagnosed group, the "Conners Parent Rating Scale - Revised Short" and "Conners Teacher Rating Scale - Revised Short" will be applied to determine the severity of the disorder, symptoms, and predominant subtyping. After the diagnosis is made and evaluated according to the exclusion criteria, blood samples will be taken from the patient after a 10-12 hour fasting period, between 9-12 AM, in a yellow-capped tube, before the routine methylphenidate treatment is used. After waiting for 10-20 minutes at room temperature, the sample will be centrifuged at 3000 RPM for 20 minutes, and the serum will be collected in Eppendorf tubes and stored at -80°C until analysis. After 3 months of treatment, blood samples will be taken again in the same manner and stored. Once all the samples are collected, the serum samples will be analyzed for total antioxidant status (TAS), total oxidant status (TOS), malondialdehyde (MDA), superoxide dismutase (SOD), and oxidized LDL levels according to the human ELISA kit protocols at the Biochemistry Laboratory of Bakırköy Dr. Sadi Konuk Training and Research Hospital by biochemist Dr. Hacer Eroğlu İçli. After 3 months of treatment, the Conners Parent Rating Scale - Revised Short and Conners Teacher Rating Scale - Revised Short forms will be applied again. In addition to the markers, the Oxidative Stress Index (OSI = TOS/TAS) will be calculated and included in the evaluation before and 3 months after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* - A diagnosis of "Attention Deficit Hyperactivity Disorder" according to DSM-5 TR, and the initiation or planned initiation of methylphenidate treatment as part of routine care.
* Being between the ages of 6 and 11.
* Providing consent to participate in the study after being informed about the study.

Exclusion Criteria:

* - Presence of a psychiatric disorder diagnosis other than "Attention Deficit Hyperactivity Disorder."
* The diagnosis of "Attention Deficit Hyperactivity Disorder" has been made, but methylphenidate treatment has not been planned.
* Being under the age of 6 or over the age of 11.
* Presence of organic brain damage, mental retardation, autism spectrum disorder, neurological diseases, or any physical illness affecting neurocognitive functions.
* A history of alcohol and/or psychoactive substance use.
* Presence of ongoing active infection, allergic diseases, or chronic illness.
* Previous use of psychiatric medication.
* Presence of a chronic illness.
* Use of regular medication.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Patients who applied to Bakırköy Prof. Dr. Mazhar Osman Mental Health and Neurological Diseases Training and Research Hospital, diagnosed with Attention Deficit Hyperactivity Disorder, deemed suitable for methylphenidate treatment, and for whom methylphenidate treatment is planned, have been referred to us.
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2024-06-26 (Actual); Primary Completion 2025-01-06 (Actual); Study Completion 2025-01-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Bakırköy Prof. Dr. Mazhar Osman Mental Health and Neurological Diseases Training and Research Hospital, Istanbul, Bakirkoy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The participants' age, scores of the clinical scales examined in the study, and levels of serum samples will be shared. In other words, the necessary data relevant to the purpose of the study will be shared.
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] Smaga I, Niedzielska E, Gawlik M, Moniczewski A, Krzek J, Przegalinski E, Pera J, Filip M. Oxidative stress as an etiological factor and a potential treatment target of psychiatric disorders. Part 2. Depression, anxiety, schizophrenia and autism. Pharmacol Rep. 2015 Jun;67(3):569-80. doi: 10.1016/j.pharep.2014.12.015. Epub 2015 Jan 5. PMID 25933971
- [Result] Koc S, Guler EM, Derin S, Gultekin F, Aktas S. Oxidative and Inflammatory Parameters in Children and Adolescents With ADHD. J Atten Disord. 2023 Jun;27(8):880-886. doi: 10.1177/10870547231159907. Epub 2023 Mar 6. PMID 36879528
- [Result] Corona JC. Role of Oxidative Stress and Neuroinflammation in Attention-Deficit/Hyperactivity Disorder. Antioxidants (Basel). 2020 Oct 23;9(11):1039. doi: 10.3390/antiox9111039. PMID 33114154
- [Result] Kul M, Unal F, Kandemir H, Sarkarati B, Kilinc K, Kandemir SB. Evaluation of Oxidative Metabolism in Child and Adolescent Patients with Attention Deficit Hyperactivity Disorder. Psychiatry Investig. 2015 Jul;12(3):361-6. doi: 10.4306/pi.2015.12.3.361. Epub 2015 Jul 6. PMID 26207130
- [Result] Cunill R, Castells X. [Attention deficit hyperactivity disorder]. Med Clin (Barc). 2015 Apr 20;144(8):370-5. doi: 10.1016/j.medcli.2014.02.025. Epub 2014 Apr 29. Spanish. PMID 24787685
- [Result] Leung AK, Hon KL. Attention-Deficit/Hyperactivity Disorder. Adv Pediatr. 2016 Aug;63(1):255-80. doi: 10.1016/j.yapd.2016.04.017. No abstract available. PMID 27426904

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Initially, 39 patients were enrolled in the study, and each patient who dropped out of the study during follow-up was replaced by a new patient in accordance with the protocol. Thus, a total of 53 patients were included in the study and 14 patients left the study for various reasons.
Groups:
- Patients Diagnosed With Attention Deficit Hyperactivity: Patients diagnosed with attention deficit hyperactivity and planned to start methylphenidate treatment
Period: Overall Study
Arm/Group | Patients Diagnosed With Attention Deficit Hyperactivity
Started | 53
Completed | 39
Not Completed | 14
Not completed — Lost to Follow-up | 5
Not completed — stigmatization concerns | 2
Not completed — medication refusal | 2
Not completed — concerns about possible side effects | 2
Not completed — wanting to seek another specialist opinion | 2
Not completed — side effects (dizziness) | 1

BASELINE CHARACTERISTICS:
Arm/Group | Patients Diagnosed With Attention Deficit Hyperactivity
Number analyzed (Participants) | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.38 (1.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Turkey | 39
Body Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 27.95 (7.38)
body mass index (BMI) [Mean (Standard Deviation); unit: kilogram(kg)/height(metre)²] | 16.60 (1.96)

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Oxidant Status
Description: Total Oxidant Status (TOS) level was measured according to the human ELISA kit protocol. Serum samples from 39 patients were compared immediately before and after 3 months of treatment. TOS was measured according to the human ELISA kit protocol as follows (bioassay technology laboratory, Cat.No E1599Hu):
  Standards added to wells. 40μl of serum sample was added to the sample wells, followed by 10μl of anti-TOS antibody. Incubated at 37°C for 60 minutes. plate was washed 5 times with wash buffer. 50μl of substrate solution A was added to the wells and then 50μl of substrate solution B was added to each well. The plate was incubated for 10 minutes at 37°C in the dark. 50μl of Stop Solution was added to the wells and the blue color immediately changed to yellow. The optical density (OD value) of each well was determined using a microplate reader set to 450 nm within 10 min after adding the stop solution.
Time Frame: Immediately before starting the treatment and up to the 3rd month of treatment.
Measure: Mean (Standard Deviation); unit: U/ml
Groups:
- Patients Diagnosed With Attention Deficit Hyperactivity: Children aged 6 to 11 years with attention deficit hyperactivity
Arm/Group | Patients Diagnosed With Attention Deficit Hyperactivity
Number analyzed (Participants) | 39
U/ml
  total oxidant status (before starting treatment) | 6.29 (5.37)
  total oxidant status (after starting treatment) | 5.62 (4.76)
Statistical Analysis 1: Comparison: Patients Diagnosed With Attention Deficit Hyperactivity; Test type: Superiority; p < 0.001, t-test, 2 sided; paired t-test

2. Primary Outcome: Change in Total Antioxidant Status
Description: Total antioxidant status (TAS) level was measured according to the human ELISA kit protocol. Serum samples from 39 patients were compared immediately before and after 3 months of treatment.TAS was measured according to the human ELISA kit protocol as follows (bioassay technology laboratory, Cat.No E4350Hu):
  Standards added to wells. 40μl of serum sample was added to the sample wells, followed by 10μl of anti-TOS antibody. Incubated at 37°C for 60 minutes. plate was washed 5 times with wash buffer. 50μl of substrate solution A was added to the wells and then 50μl of substrate solution B was added to each well. The plate was incubated for 10 minutes at 37°C in the dark. 50μl of Stop Solution was added to the wells and the blue color immediately changed to yellow. The optical density (OD value) of each well was determined using a microplate reader set to 450 nm within 10 min after adding the stop solution.
Time Frame: Immediately before starting the treatment and up to the 3rd month of treatment.
Measure: Mean (Standard Deviation); unit: U/ml
Arm/Group | Patients Diagnosed With Attention Deficit Hyperactivity
Number analyzed (Participants) | 39
U/ml
  total antioxidant status (before starting treatment) | 7.79 (5.65)
  total antioxidant status (after starting treatment) | 7.33 (5.40)
Statistical Analysis 1: Comparison: Patients Diagnosed With Attention Deficit Hyperactivity; Test type: Superiority; p = 0.021, t-test, 2 sided; paired t-test

3. Primary Outcome: Change in Superoxide Dismutas
Description: superoxide dismutas level was measured according to the human ELISA kit protocol. Serum samples from 39 patients were compared immediately before and after 3 months of treatment. Superoxide dismutas was measured according to the human ELISA kit protocol as follows (bioassay technology laboratory, Cat.No E0918Hu): Standards added to wells. 40μl of serum sample was added to the sample wells, followed by 10μl of anti-TOS antibody. Incubated at 37°C for 60 minutes. plate was washed 5 times with wash buffer. 50μl of substrate solution A was added to the wells and then 50μl of substrate solution B was added to each well. The plate was incubated for 10 minutes at 37°C in the dark. 50μl of Stop Solution was added to the wells and the blue color immediately changed to yellow. The optical density (OD value) of each well was determined using a microplate reader set to 450 nm within 10 min after adding the stop solution.
Time Frame: Immediately before starting the treatment and up to the 3rd month of treatment.
Population: 2 patients were excluded because there was no reaction and no color change in the measurement.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Patients Diagnosed With Attention Deficit Hyperactivity
Number analyzed (Participants) | 37
U/L
  superoxide dismutas (before starting treatment | 175.89 (158.95)
  superoxide dismutas (after starting treatment) | 160.88 (143.49)
Statistical Analysis 1: Comparison: Patients Diagnosed With Attention Deficit Hyperactivity; Test type: Superiority; p = 0.003, t-test, 2 sided; paired t-test

4. Primary Outcome: Change in Malondialdehyde
Description: Malondialdehyde (MDA) level was measured according to the human ELISA kit protocol. Serum samples from 39 patients were compared immediately before and after 3 months of treatment. MDA was measured according to the human ELISA kit protocol as follows (bioassay technology laboratory, Cat.No E1371Hu):
  Standards added to wells. 40μl of serum sample was added to the sample wells, followed by 10μl of anti-TOS antibody. Incubated at 37°C for 60 minutes. plate was washed 5 times with wash buffer. 50μl of substrate solution A was added to the wells and then 50μl of substrate solution B was added to each well. The plate was incubated for 10 minutes at 37°C in the dark. 50μl of Stop Solution was added to the wells and the blue color immediately changed to yellow. The optical density (OD value) of each well was determined using a microplate reader set to 450 nm within 10 min after adding the stop solution.
Time Frame: Immediately before starting the treatment and up to the 3rd month of treatment.
Measure: Median (Inter-Quartile Range); unit: nmol/ml
Arm/Group | Patients Diagnosed With Attention Deficit Hyperactivity
Number analyzed (Participants) | 39
nmol/ml
  Malondialdehyde (before starting treatment) | 9.58 [7.35 to 9.94]
  Malondialdehyde (after starting treatment) | 8.65 [7.00 to 13.61]
Statistical Analysis 1: Comparison: Patients Diagnosed With Attention Deficit Hyperactivity; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)

5. Primary Outcome: Change in Ox-LDL
Description: Ox-LDL level was measured according to the human ELISA kit protocol. Serum samples from 39 patients were compared immediately before and after 3 months of treatment. Ox-LDL was measured according to the human ELISA kit protocol as follows (bioassay technology laboratory, Cat.No E1521Hu):
  Standards added to wells. 40μl of serum sample was added to the sample wells, followed by 10μl of anti-TOS antibody. Incubated at 37°C for 60 minutes. plate was washed 5 times with wash buffer. 50μl of substrate solution A was added to the wells and then 50μl of substrate solution B was added to each well. The plate was incubated for 10 minutes at 37°C in the dark. 50μl of Stop Solution was added to the wells and the blue color immediately changed to yellow. The optical density (OD value) of each well was determined using a microplate reader set to 450 nm within 10 min after adding the stop solution.
Time Frame: Immediately before starting the treatment and up to the 3rd month of treatment.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Patients Diagnosed With Attention Deficit Hyperactivity
Number analyzed (Participants) | 39
ng/mL
  Ox-LDL (before starting treatment) | 34.19 [26.36 to 60.96]
  Ox-LDL (after starting treatment) | 29.59 [25.24 to 56.67]
Statistical Analysis 1: Comparison: Patients Diagnosed With Attention Deficit Hyperactivity; Test type: Superiority; p = 0.001, Wilcoxon (Mann-Whitney)

6. Primary Outcome: Change in Oxidative Stress Index (OSI)
Description: Oxidative Stress Index (OSI) level was measured according to the human ELISA kit protocol. Serum samples from 39 patients were compared immediately before and after 3 months of treatment.
  OSI is an index created by the ratio of TOS to TAS. OSI is a parameter that shows the direction in which the body's oxidative stress balance shifts. An increase or decrease in the OSI value indicates that the oxidative balance has changed. While an increase in OSI value indicates a change in balance in favor of oxidants; a decrease in OSI value indicates a change in balance in favor of anti-oxidants.
Time Frame: Immediately before starting the treatment and up to the 3rd month of treatment.
Measure: Mean (Standard Deviation); unit: Index
Arm/Group | Patients Diagnosed With Attention Deficit Hyperactivity
Number analyzed (Participants) | 39
Index
  Oxidative Stress Index (OSI) (before starting treatment) | 0.75 (0.12)
  Oxidative Stress Index (OSI) (after starting treatment) | 0.72 (0.12)

ADVERSE EVENTS:
Time Frame: 3 months
Description: Patients diagnosed with attention deficit hyperactivity and planned to receive methylphenidate treatment were included in the study. Patients eligible for methylphenidate treatment due to indication were included. Therefore, there were no patients at risk of death or serious adverse events.
Arm/Group | Patients Diagnosed With Attention Deficit Hyperactivity
All-Cause Mortality (participants affected / at risk) | 0/53
Serious Adverse Events (participants affected / at risk) | 0/53
Other Adverse Events (participants affected / at risk) | 26/53
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients Diagnosed With Attention Deficit Hyperactivity (N=53)
loss of appetite (General disorders) | 20 — In 8 children, this side effect disappeared at 3-month follow-up. In 12 children, this side effect persisted for 3 months.
abdominal pain (temporary) (General disorders) | 5
headache (temporary) (General disorders) | 3
nausea (temporary) (General disorders) | 5
stagnation (temporary) (General disorders) | 6
weight loss (General disorders) | 3 — In 1 child, this side effect disappeared at 3 months follow-up. In 2 children, this side effect persisted for 3 months.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-03-18): https://cdn.clinicaltrials.gov/large-docs/12/NCT06844812/Prot_SAP_ICF_001.pdf